CLINICAL TRIAL: NCT06932302
Title: At-Home Neuromodulation for Female Sexual Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Timothy Bruns, Associate Professor of Biomedical Engineering, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00265573
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Female Sexual Dysfunction
Keywords: dorsal genital nerve stimulation; neuromodulation
MeSH Terms: interventions — Electric Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Nerve Stimulation only (Experimental): Pre-menopausal women and post-menopausal women will be recruited. Individuals in this group will only perform dorsal genital nerve stimulation.
  Interventions: Device: Electrical Stimulation
- Nerve Stimulation and Vibration (Experimental): Pre-menopausal women and post-menopausal women will be recruited. Individuals in this group will perform dorsal genital nerve stimulation and use a smart vibrator.
  Interventions: Device: Electrical Stimulation; Device: Smart vibrator
- Vibration only (Active Comparator): Pre-menopausal women and post-menopausal women will be recruited. Individuals in this group will only use a smart vibrator.
  Interventions: Device: Smart vibrator

INTERVENTIONS:
Device: Electrical Stimulation — Electrical stimulation of the dorsal genital nerve will be accomplished using the UCon system and patch electrodes developed by InnoCon. The UCon system includes a programmable control unit; leads that connect to the control unit and electrodes; a silicone surface electrode; a reference electrode; and a remote control for quick on and off toggling of stimulation.
  Other Names: UCon patch system
  Arms: Nerve Stimulation and Vibration; Nerve Stimulation only
Device: Smart vibrator — Subjects will use a smart vibrator at home twice a week during the study. The Lioness smart vibrator records physiological responses during use.
  Arms: Nerve Stimulation and Vibration; Vibration only

SUMMARY:
This pilot study investigates the regular use of non-invasive dorsal genital nerve stimulation (DGS) for the treatment of female sexual dysfunction (FSD). The researchers aim to determine whether subjects with FSD can correctly follow an at-home treatment regimen and to demonstrate that DGS can improve FSD arousal symptoms in premenopausal and postmenopausal women. Some subjects will use a smart vibrator for comparison to DGS.

ELIGIBILITY:
Inclusion Criteria:

* Capable of speaking and understanding English.
* Able to comprehend the clinical study procedures and provide informed consent.
* Identified as having female sexual dysfunction with a Female Sexual Function Index (FSFI) score of 26.55 or less and a score of 3 or less on one or more of the FSFI subdomains of lubrication, arousal, and orgasm.
* Willing and able to adhere to the study protocol
* Able to attend experimental sessions at Michigan Medicine at both the start and conclusion of the study.

Exclusion Criteria:

* Not currently sexually active.
* Pregnant or planning to get pregnant during the study period.
* History of a neurological disorder or impairments affecting pelvic organ function, including diagnosed with dorsal genital nerve damage, lower motor dysfunction, or other related conditions.
* Implanted with a neurostimulator for bladder or bowel function.
* Have a skin condition that would predispose them to sensitivity to the stimulation electrodes.
* Female sexual dysfunction limited solely to low desire, without issues in lubrication, arousal, or orgasm.
* Clinically diagnosed bladder dysfunction, pelvic pain, or other pelvic organ symptoms; or a score of 8 or higher on the American Urological Association Symptom Index (AUASI).
* Unable or unwilling to adhere to the study protocol
* Simultaneously participating in another research study that may affect the results of this study.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Number of dorsal genital nerve stimulation (DGS) sessions performed | Approximately day 22
Number of related adverse events | Up to week 9
  Study-related AEs include incidents such as device zapping, skin irritation, back cramps, or falls due to sitting for 30 minutes of stimulation.

SECONDARY OUTCOMES:
Change in Female Sexual Function Index (FSFI) total scores | Baseline and approximately day 22
  The FSFI is a 19-question survey assessing sexual function in 6 different domains (desire, arousal, lubrication, orgasm, satisfaction, and pain). Each question asks subjects to rate an aspect of their sexual function on a scale from 0 or 1 to 5, depending on the question. The total score for each subdomain is multiplied by a factor so that the maximum score is 6. The total score is out of 36, with the cutoff score for overall dysfunction being 26.55. Subdomain scores of 3 or less indicate dysfunction in the respective subdomain. The FSFI will be conducted before the first study visit and again within one week after completion of the at-home stimulation period in order to see if scores have changed over the course of the treatment.
The Patient Global Impression of Change (PGIC) survey score | Up to week 9
  The Patient Global Impression of Change (PGIC) is a 1-question survey asking patients to describe the change in their condition with a number from 1 to 7. Each number is paired with a description, where 1 represents "No change (or condition is worse)" and 7 represents "A great deal better, and a considerable improvement that has made all the difference". The PGIC will be administered within one week after completion of at-home stimulation, and again 1 month later in order to assess the patient's perception of their change in symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Bruns, PhD, Principal Investigator — University of Michigan; Priyanka Gupta, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No